CLINICAL TRIAL: NCT00479271
Title: The Dementia Home Care Project: a Randomised Controlled Trial to Evaluate the Effectiveness of a Home Care Program for Supporting Caregivers of Persons With Dementia in Developing Countries: a Randomised Controlled Trial From Goa, India
Brief Title: Evaluating the Effectiveness of a Community Based Intervention for Persons With Dementia and Their Caregivers in a Developing Country
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: The Dementia Society of Goa, India (Other); Goa Medical College (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: DSG001
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2007-05

CONDITIONS: Dementia; Behavioral Symptoms; Mental Health
Keywords: RCT; Dementia; community trial; Homebased care; caregiver burden; Behavioural problems; Dementia in subjects; behavioral problems in subjects; Mental health of carers
MeSH Terms: conditions — Dementia; Behavioral Symptoms; Psychological Well-Being; Caregiver Burden; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home Care (Active Comparator): A flexible home-care program tailored to the needs of the individual and the family. The components of the intervention will include:
  1. Basic education about dementia (what is the disease, its course, its features etc)
  2. Education about common behaviour problems and how they can be managed
  3. Support to the carer, for example for an elderly carer living alone with the patient, in activities of daily living
  4. Referral to specialists when behaviour problems are severe and warrant medication intervention (sedatives).
  Interventions: Behavioral: Home based, flexible, stepped care intervention
- Wait-list (Other): This group will be put on a waiting list to receive the intervention after 6 months. Families will be free to choose any health care they desire during the waiting period.
  Interventions: Behavioral: Home based, flexible, stepped care intervention after 6 months. Families will be free to choose any health care they desire during the waiting period.

INTERVENTIONS:
Behavioral: Home based, flexible, stepped care intervention — Home based, flexible, stepped care intervention
  Arms: Home Care
Behavioral: Home based, flexible, stepped care intervention after 6 months. Families will be free to choose any health care they desire during the waiting period. — Home based, flexible, stepped care intervention after 6 months. Families will be free to choose any health care they desire during the waiting period.
  Arms: Wait-list

SUMMARY:
The aim of this trial was to apply a home based, flexible, stepped-care intervention designed to improve the awareness and knowledge of family caregivers regarding dementia, to maximise their caregiving resources and to improve their caregiving skills. A Randomized Controlled Trial (RCT) will be used to evaluate the same wherein the intervention group will get the services immediately and the control arm would receive the same after a period of 6 months.

DETAILED DESCRIPTION:
Service development for older people with dementia in India needs to take account of the fact that dementia tends to be a hidden problem. Thus, dementia is generally perceived to be part of normal ageing, and not a health condition, and families rarely present to health services, who are generally ignorant of most cases in their community. Health services are often ill-equipped to meet the needs of older persons. Health care, even primary care, is clinic-based; the older person must attend the clinic or hospital, often involving a long journey and waiting time. The assessment and treatment that they receive is orientated towards acute rather than chronic conditions. Thus, home-based interventions provide a practical alternative to clinic-based interventions for persons affected by dementia.

The probable cases of dementia will be identified with the help of key informants (doctors, priests, health workers, local leaders) in two of the most populated talukas of Goa (Bardez and Tiswadi,). All probable cases will be examined by a trained clinician to confirm the diagnosis of dementia. Cases will be randomized to receive the intervention or placed in a waiting list group who will receive the intervention after 6 months. The intervention will be delivered by a trained community Home Care Advisors (HCA), supported when required by the Principal Investigators and clinical consultants. The principal outcomes being evaluated are carer burden and mental health, behavioral problems in the person with dementia, and costs of illness.

Objectives

The project has two specific objectives:

* To adapt and apply a flexible, stepped-care intervention designed to improve the awareness and knowledge of family caregivers regarding dementia, to maximise their caregiving resources and to improve their caregiving skills.
* To evaluate the efficacy and cost-effectiveness of the intervention in reducing carer burden, improving behaviour problems in elderly persons with dementia and reducing the costs of illness.

The intervention is designed to provide family caregivers with information about dementia syndrome, assistance in setting up local support groups with other caregivers, and training in strategies to better manage common behavioural problems in the home setting. This package would form the basis of the community intervention to be delivered in the proposed project. The third group of carers are medical personnel. Some patients with dementia suffer from behavioural or psychiatric problems which may improve considerably with the judicious use of psychotropic medication. The use of such medication requires the assessment and evaluation by a physician who has had basic training in the use of sedative medication in elderly people.

Baseline interview:

The baseline assessment of the demographic characteristics of the family, the background information about the Principal carer and the subject, costs of caring for the person with dementia, behavioural problems in the subject, perceived burden and the impact on the carers mental health. This information will be made available to the HCAs before they initiate the intervention.

Randomisation and Intervention: All subjects will be allocated a study number and randomised into two groups by a person at the central office. The person involved with the process of randomization will be blind to the status of the subject. Random number table will be used for the process. The HCA will then be informed of the family allotted to them for intervention.

After randomization the families will be divided into the following two groups:

Intervention and control

The medical intervention followed a treatment protocol.

Intervention

Following suitable training, the Home Care Advisors will apply a flexible home-care program tailored to the needs of the individual and the family. The components of the intervention will include:

* Basic education about dementia (what is the disease, its course, its features etc)
* Education about common behaviour problems and how they can be managed
* Support to the carer, for example for an elderly carer living alone with the patient, in activities of daily living
* Referral to specialists when behaviour problems are severe and warrant medication intervention (sedatives).

Instruments used for evaluation:

* Socio demographic characteristics of the person with dementia and the caregiver
* Everyday Abilities Scale for India (EASI): This questionnaire consisting of 12 questions, has been developed and widely used to test the functional abilities of daily living relevant to Indian subjects[11]
* Neuro-Psychiatric Inventory (NPI) Questionnaire: This instrument consists of two parts; the first measures the severity of the problem behaviours associated with the condition on a scale of 1-3 (NPI- S); the second measures the perceived distress of the problem behaviours by the caregiver on a scale of 0-5 (NPI -D)[12].
* Zarit Burden scale (ZBS): This is the most widely used scale in the studies of caregiver burden and encompasses the physical, emotional and financial burden as perceived by the caregiver[13].
* General Health Questionnaire (GHQ): The 12 question GHQ is used to measure the psychological impact on the caregivers' mental health.

Control Group This group will be put on a waiting list to receive the intervention after 6 months. Families will be free to choose any health care they desire during the waiting period.

The broad outlines for the sessions for the intervention are as follows:

Understanding the Family Support system:

In this session the Home Care Advisor ( HCA ) will try and identify the principal carer, the family structure and the pattern of informal care provided to the person with dementia. They will try and identify stressors in the family like unemployment, alcoholism, financial constraints, etc. They will try to understand the possible ways to restructure the informal support system if required.

Explaining what is Dementia :

This session will first begin with accessing the carer's knowledge about the disease and help the carer understand the diagnosis and prognosis. The HCA will also give the family an overall idea of the prevalence of the disorder in the community.

Identifying and managing caregiver burnout:

The success of the stepped care model depends on identifying the stress in the carer and help them effectively manage it. A carer who is emotionally disturbed will not be in a position to gain new knowledge or learn new skills. In a nuclear family the caregiver is most likely to be the daughter in law who will have a number of other responsibilities which she carries out at the cost of her mental and physical health. Over the years her role becomes a routine and often a thankless job. The HCAs will try and create an environment which is supportive and sensitive to the needs of the carer.

Stress Management and Relaxation:

During this session the HCA will train the carer in stress management and relaxation techniques. If the non pharmacological methods do not work, they will advise and arrange for a visit to a psychiatrist for appropriate management.

Managing Problem Behaviours:

In this session the HCA will try and identify the problem behaviours like wandering, repetitive behaviours, hallucinations, screaming episodes, clinging, incontinence etc. They will help carers understand them and provide practical tips on management of problem behaviours at home. The case will be discussed with the counselor and the clinical consultants for their inputs.

Structuring a Day:

The HCA will give the carer tips on how to structure a day so as to make it easier for the subject and the carer to manage time and adjust to the changes taking place.

Nutrition:

Nutrition is often the major concern of the carers. The HCA will advise the carer on how to improve the nutrition of the subject and the family.

Management of Associated Disorders:

The Home Care advisors will be equipped with knowledge on the ailments that the person with dementia is likely to have. The subject being old may have a number of disorders like Diabetes Mellitus, Hypertension, Ischemic Heart Disease, renal failure which are neglected as the disease progresses. The Home Care Advisors will try and find out if any of these conditions exist and advise the appropriate referral for the management so as to improve the quality of life.

Meeting with the Clinical Consultants and Counselor; The Home Care Advisors will meet the clinical consultants every week to discuss the progress of the case and the arrange for a visit whenever required. The Clinical consultants will also provide the appropriate advise for the management of the subject. They will meet the counselor every fortnightly to discuss the social and emotional aspects of the intervention.

Networking:

The HCAs will try and arrange a meeting of the carers and encourage them share their experiences with each other. Group sessions, film shows and lectures will be arranged at the meeting. They will be encouraged to meet and form support groups.

ELIGIBILITY:
Inclusion Criteria:

* All probable cases will be examined by a trained clinician (AD) to confirm the diagnosis of dementia according to DSM IV criteria and graded using the Clinical Dementia Rating (CDR) Scale.
* CDR mild and moderate dementia.
* The principal caregiver, as identified by the family, was enrolled for the trial. The principal caregiver was generally the spouse, although in some instances another family member was the principal caregiver, particularly when the spouse was not in a position to care.

Exclusion Criteria:

* CDR severe dementia or severe co-morbid physical health conditions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure(s) evaluate the efficacy and cost-effectiveness of the intervention in reducing carer burden, improving behaviour problems in elderly persons with dementia and reducing the costs of illness. | by the end of the study

SECONDARY OUTCOMES:
Measure the service requirements, average number of visits by Home Care Advisor, visits by Psychiatrists, need for medication, effect of intervention on survival and overall quality of life of the person with dementia as well as the carer | by the end of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Patel, Principal Investigator — London School of Hygiene and Tropical Medicine; Amit Dias, MD,DGM,DTM&H, Principal Investigator — The Dementia Society of Goa, & Goa Medical College
Locations (1):
- The Dementia Society of Goa, Porvorim, Goa, India

REFERENCES:
- [Derived] Dias A, Dewey ME, D'Souza J, Dhume R, Motghare DD, Shaji KS, Menon R, Prince M, Patel V. The effectiveness of a home care program for supporting caregivers of persons with dementia in developing countries: a randomised controlled trial from Goa, India. PLoS One. 2008 Jun 4;3(6):e2333. doi: 10.1371/journal.pone.0002333. PMID 18523642